CLINICAL TRIAL: NCT02745210
Title: Non-invasive Clinical Imaging of Cerebral Metabolism Following Brain Injury Using 13C Magnetic Resonance Spectroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The acquisition sequence was incompatible with MRI hardware
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Brenda Bartnik Olson, PhD, Principal Investigator, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 59093
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): 13C Magnetic resonance (MR) spectroscopy.
  Interventions: Diagnostic Test: 13C magnetic resonance spectroscopy

INTERVENTIONS:
Diagnostic Test: 13C magnetic resonance spectroscopy — acquisition of 13C MR spectroscopy in the brain
  Other Names: 13C MRS

SUMMARY:
Despite the decline in fatal traumatic brain injury (TBI) incidence in recent years, TBI morbidity remains a public health challenge and is the leading cause of disability in the United States. Detailed knowledge of the metabolic alterations following TBI will provide a significant advancement to our understanding of the hypometabolic response to TBI, which is key information for the future development and testing of novel therapeutic interventions that by-pass or compensate for the metabolic dysfunction.

The goal of this study is to determine the clinical utility of in vivo 13C MRS to identify specific metabolic alterations following TBI. We hypothesize that following TBI, metabolic pathways are altered causing an incomplete oxidative of glucose in neurons and astrocytes resulting in a decrease in cerebral metabolism.

DETAILED DESCRIPTION:
Despite the decline in fatal traumatic brain injury (TBI) incidence in recent years, TBI morbidity remains a public health challenge and is the leading cause of disability in the United States To combat these effects, new research is needed to identify mechanisms of injury that will lead to potential targets for therapeutic interventions that improve neurological outcome. One promising area of research is the cerebral metabolic dysfunction following TBI. Studies of post-traumatic cerebral metabolism have shown that cerebral metabolic rate of glucose (CMRglc) decreases for a period of days, weeks or months after injury with the duration and degree of hypometabolism correlating to level of consciousness and a strong predictor of long-term neurological outcome. However, specific changes in intermediary carbohydrate metabolic pathways have not yet been identified. In addition, the role of astrocyte metabolism in the post-injury metabolism has not been studied. This study uses in vivo 13C magnetic resonance spectroscopy (MRS) at 3 Tesla, a novel method in the clinical study of TBI, to non-invasively study the metabolic fate and flux of glucose (metabolized in both neurons and astrocytes) and acetate (metabolized in astrocytes) through metabolic pathways during the hypometabolic period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be at least 18 years of age without gender or ethnic restrictions.
2. Severe accidental TBI defined as the lowest post-resuscitation GCS < 8 prior to administration of sedatives or paralytics.
3. Eligibility for MRI per routine screening checklist.

Exclusion Criteria:

1. History of neurosurgical intervention, excluding the placement of ventriculostomy shunt
2. History of a prior known brain injury with associated loss of consciousness.
3. History of a known neurological disorder prior to qualifying injury.
4. History of psychiatric disorder.
5. History of diabetes or current unstable serum glucose level.
6. Renal insufficiency or known history of kidney disease.
7. Known contraindication to MRI such as, pacemaker, pregnancy, and/or other non-MR compatible implanted device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from medical, surgical, or neurological services of LLUMC. Non-injured participants were recruited from MRI staff, Loma Linda University student or Resident populations
Groups:
- Traumatic Brain Injury: Participants with TBI undergoing 13C Magnetic resonance (MR) spectroscopy.
- Control: control (non-injured) participants undergoing 13C Magnetic resonance (MR) spectroscopy.
Period: Overall Study
Arm/Group | Traumatic Brain Injury | Control
Started | 0 | 9
Completed | 0 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No traumatic brain injury participants were recruited
Groups:
- Total: Total of all reporting groups
Arm/Group | Traumatic Brain Injury | Control | Total
Number analyzed (Participants) | 0 | 9 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 33 (7.71) | 33 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 0 | 4 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Detection of 13C Enriched Cerebral Metabolites
Description: Direct detection, localized in vivo 13C MRS will be used to measure the 13C enrichment of glutamate and glutamine following an infusion of 30% isotopically enriched [1-13C] glucose and [1, 2-13C2] acetate.
Time Frame: 5 years
Population: We were not successful in out attempt to collect localized in vivo 13C MRS thus there were no metabolite enrichments to measure and include in the measure data table.
Arm/Group | Experimental
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse event collection was based on self-reporting by participants
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT02745210/Prot_SAP_000.pdf